CLINICAL TRIAL: NCT01261234
Title: Effect of Cilostazol on In-stent Restenosis After Carotid Artery Stenting; Multi-center, Prospective, Randomized, Open-label Blind-endpoint Trial
Brief Title: Carotid Artery Stenting With Cilostazol Addition for Restenosis
Acronym: CAS-CARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kobe City General Hospital (Other)
Collaborators: Chiba University (Other); Nagoya University (Other); Mie University (Other); Wakayama Medical University (Other); Kyoto University (Other); Osaka University (Other); Kobe University (Industry); Foundation for Biomedical Research and Innovation (Other); Okayama University (Other); Yamaguchi University Hospital (Other); Fukuoka University (Other); Nagasaki University (Other)
Responsible Party: Principal Investigator, Nobuyuki Sakai, Director, Neurosurgery, Kobe City General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TRIBRAIN1010; UMIN000004705 (Other: University hospital Medical Information Network, Japan)
Record Dates: First submitted 2010-12-11; First posted 2010-12-16 (Estimated); Last update posted 2019-10-16 (Actual); Status verified 2019-10

CONDITIONS: In-stent Restenosis After Carotid Artery Stenting
Keywords: Carotid Artery Disease; Carotid Artery Stenting; In stent restenosis; Cardiovascular event; Intima Media Thickness
MeSH Terms: conditions — Carotid Artery Diseases | interventions — Cilostazol; Population Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cilostazol group (Experimental): Continuous administration of cilostazol (unrestricted use of other antiplatelet agents and concomitant drugs)
  Interventions: Drug: Cilostazol or Non-Cilostazol
- Non-Cilostazol group (Active Comparator): Antiplatelet agent other than cilostazol (unrestricted use of concomitant drugs)
  Interventions: Drug: Cilostazol or Non-Cilostazol

INTERVENTIONS:
Drug: Cilostazol or Non-Cilostazol — Cilostazol group administrate 100-200mg/day per oral, unrestricted use of other antiplatelet agents and concomitant drugs.
  Other Names: Cilostazol (Pretal) group; Non-Cilostazol (Pretal) group

SUMMARY:
CAS-CARE study was conducted to evaluate the inhibitory effect of cilostazol, compared to that of other antiplatelet drugs, on in-stent restenosis following carotid artery stenting (CAS) in patients scheduled to undergo CAS. Study design is Multicenter Prospective Ranodomized Controlled Study, rondomized by cilostazol/non-cilostazol group prior to CAS. 900 patients will be enrolled for 2 years and followed 2 years with in-stent restenosis after CAS, evaluated by carotid ultrasound and angiography.

DETAILED DESCRIPTION:
Restenosis after carotid artery stenting (CAS) is a critical issue. Cilostazol can reduce restenosis after interventions in coronary or femoropopliteal arteries. The investigators confirmed and published periprocedural cilostazol administration reduced incidences of in-stent restenosis (ISR) or target vessel revascularization (TVR) after CAS, retrospectively.

CAS-CARE study is Multicenter Prospective Ranodomized Controlled Study. Patients, scheduled for CAS within 30 days, 50% or more symptomatic carotid stenosis or 80% or more asymptomatic carotid stenosis, will enroll and randomize by cilostazol/non-cilostazol group. 900 patients will be enrolled for 2 years and followed 2 years with in-stent restenosis after CAS, evaluated by carotid ultrasound and angiography. And, evaluate cardiovascular events, including stroke, myocardial infarction, and hemorrhagic events in periprocedural period and followed period. In this study, ISR is diagnosed by ultrasound and DSA/CTA. Equivalence of CTA to ultrasound will be studied.

ELIGIBILITY:
Inclusion Criteria:

* 50% or more symptomatic carotid artery stenosis or 80% or more asymptomatic carotid artery stenosis
* scheduled for carotid artery stenting within 30 days
* 45 or more years-old and less than 80 years old
* antiplatelet agents can be administratered orally
* follow-up is anticipated possible for 2 years after CAS
* self-supporoted in daily activities (modified Rankin Scale 2 or less)
* patients who have given informed consent to participation in the study

Exclusion Criteria:

* received endovascular interevention
* scheduled for bilateral carotid intervention
* aortitis or cvasculitis
* congessive heart failure
* ischemic stroke within 48 hours
* hemorrhagic stroke within 90 days
* renal failure

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 707 (Actual)
Dates: Start 2010-12 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
Presence or absence of in-stent restenosis within 2 years after CAS and time to occurrence | 2 years
  Difinition of endpoint is 50% or more in-stent restenosis detected by carotid ultrasound or angiopraphy. In cases restenosis does not occur, the final observation point will be used as the final evaluation point.

SECONDARY OUTCOMES:
Cardiovascular event, death, hemorrhagic event, in-stent restenosis, new out-stent stenosis, or retreatment of stented artery within 2 yrs | 2 years
  Any events, including death, cardiovascular event(stroke, myocardial infarction), hemorrhagic event, in-stent restenosis, new out-stent stenosis, retreatment of stented artery, within 2 years
In-stent restenosis, new out-stent stenosis, or retreatment within 2 years | 2 years
  In-stent restenosis, new out-stent stenosis detected by ultrasound or CTA/DSA, or retreatment of stented artery within 2 years
hemorrhagic event within 2 years | 2 years
  hemorrhagic stroke, major hemorrhage required 2 unit or more transfusion
stroke within 2 years | 2 years
  any ischemic or hemorrhagic stroke
In-stent restenosis, new out-stent stenosis, or retreatment of stented artery, cardiovascular event, or death from any cause within 30 days | 30 days
  Any peri-procedural events; in-stent restenosis, new out-stent stenosis, or retreatment of stented artery, cardiovascular event(stroke, myocardial infarction), or death from any cause
Severe in-stent restenosis within 2 yrs | 2 yeras
  70% or more in-stent restenosis, diagnosed by ultrasound or DSA/CTA,
Change from baseline in max-IMT in both common carotid arteries | 2 years
  Intima-Media thickness of common carotid artery measured by ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Nobuyuki Sakai, MD, DMSc, Principal Investigator — Kobe City Medical Center General Hospital; Hiroshi Yamagami, MD, PhD, Principal Investigator — Kobe City Medical Center General Hospital
Locations (1):
- Kobe City Medical Center General Hospital, Kobe, Hyōgo, Japan

REFERENCES:
- [Derived] Yamagami H, Ozaki T, Ogasawara K, Nagata I, Matsumaru Y, Yoshimura S, Sasaki M, Nagatsuka K, Minematsu K, Nagai Y, Sakai C, Matsumoto Y, Ezura M, Ishihara H, Sakai N; CAS-CARE Investigators. Randomized Controlled Trial of Cilostazol Addition for In-Stent Restenosis After Carotid Artery Stenting. Stroke. 2024 Dec;55(12):2776-2785. doi: 10.1161/STROKEAHA.124.047210. Epub 2024 Nov 25. PMID 39585936